CLINICAL TRIAL: NCT02857309
Title: Cardiac Contractility Modulation (CCM) Therapy in Subjects With Medically Refractory Heart Failure: A Randomized Efficacy Study
Brief Title: Cardiac Contractility Modulation (CCM) Therapy in Subjects With Medically Refractory Heart Failure
Acronym: IMPULSE-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrolment.
Sponsor: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID_CP_OPT2013-026
Record Dates: First submitted 2016-07-20; First posted 2016-08-05 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Angiotensin Receptor Antagonists; Mineralocorticoid Receptor Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device implant (Other): Patients randomized to the treatment group will receive optimal medical therapy for heart failure. and implantation of the OPTIMIZER System.
  Interventions: Device: OPTIMIZER; Drug: Optimal medical therapy
- Optimal medical therapy (Active Comparator): Patients randomized to the control group will receive optimal medical therapy for heart failure.
  Interventions: Drug: Optimal medical therapy

INTERVENTIONS:
Device: OPTIMIZER — The OPTIMIZER System delivers non-excitatory cardiac contractility modulation (CCM) signals to the heart that are intended to influence myocardial properties in patients with chronic heart failure. The system has no pacemaker or implantable cardioverter-defibrillator (ICD) functions.
  Arms: Device implant
Drug: Optimal medical therapy — OMT using standard heart failure (HF) drugs
  Other Names: angiotensin receptor blockers; mineralocorticoid receptor antagonists; angiotensin receptor neprilysin inhibitors

SUMMARY:
The study is designed to substantiate the efficacy of Cardiac Contractility Modulation (CCM) in the heart failure population with ejection fraction ranging between 25 and 45%. The study is designed in an adaptive manner to ensure proper statistical significance and power of the primary efficacy evaluation.

DETAILED DESCRIPTION:
This study will collect efficacy data in a randomized controlled setting, including New York Heart Association (NYHA) class II and III Heart Failure population with baseline ejection fraction (EF) of 25% to 45%.

There is previous evidence related to the beneficial effect of CCM in patients with baseline ejection fraction of <35%. While patients with EF between 35% and 45% were not prospectively studied in the original clinical study initially conducted to support Conformité Européene (CE) Marking of the OPTIMIZER System, recently available data from a randomized study that included such patients show CCM to be safe and effective in this group of patients as well. Furthermore, the literature supports that this population has very similar clinical characteristics, in practice are treated with nearly the same medications, and have similar underlying mechanisms of disease compared to patients with EF <35%. CCM has been successfully used also in patients with EF greater than 35% in routine use and in the FIX-HF-5 study.

Since the system is CE marked and since the population includes patients meeting the approved indication as well as population that has shown to benefit from CCM (EF 35%-45%), the risk involved in performing such a clinical investigation seems acceptable.

The study is designed to substantiate the efficacy of CCM in heart failure patients with EFs in the range of 25%-to-45% (inclusive). This is a prospective, randomized study comparing CCM plus optimal medical therapy (OMT) (Treatment Group) to OMT alone (Control Group) over a 24 week period. The primary endpoint shall be a comparison of changes in Peak VO2, which is an established objective physiological indicator of exercise capacity which is relevant in heart failure device studies. To further improve the accuracy and objectivity of measurements, double assessment of the Peak VO2 will be performed at each of the primary time points. Tests can be performed using upright and semi-supine bicycle ergometer or using treadmill. In sites where more than one option is available, bicycle ergometer is the preferred option. Treadmill is only allowed in case no bicycle is available at the site. Each subject shall be consistently tested using the same method throughout the study. The study is designed in an adaptive manner to ensure proper statistical significance and power of the primary efficacy evaluation.

The study will collect additional (exploratory) efficacy data on the difference between the treatment group and control group in the changes over 24 weeks in predicted survival probability. To evaluate the survival probability, two established models are used: the Seattle Heart Failure Model (SHFM), and the Meta-Analysis Global Group in Chronic Heart Failure (MAGGIC) model . These models use information collected at a certain time point to predict survival probabilities over the following years. The information used for such prediction includes status of the disease (NYHA, Left Ventricular EF (LVEF)), documented medical history and co-morbidities, documented therapies and medications, and standard blood tests values.

Additionally, hospitalization data will be collected from medical records of the site and/or from any other medical records of clinics/hospitals where the patient may have been treated for a timeframe of 12 months before enrollment and until 24 weeks after the Study Start Date (SSD).

ELIGIBILITY:
Inclusion Criteria:

* Baseline ejection fraction ≥ 25% and ≤45% (as assessed by the site)
* NYHA class II or III (chronic, not transient, heart failure) despite receiving optimal medical therapy for heart failure
* Stable medication for heart failure for at least 30 days based on patient's medical records
* Baseline Peak VO2 ≥ 10 and ≤ 18.5 ml O2/Kg/min (as assessed by the site)

Exclusion Criteria:

* Potentially correctible cause of HF (valvular, congenital, or untreated ischemic heart disease)
* Clinically significant angina pectoris
* Hospitalization for HF requiring the use of inotropic support or IV diuretics within 30 days of enrollment
* PR interval greater than 375 ms
* Permanent or persistent atrial fibrillation/flutter or cardioversion within 30 days of enrollment.
* Exercise tolerance limited by condition other than heart failure (e.g., angina, chronic obstructive pulmonary disease (COPD), peripheral vascular disease, orthopedic or rheumatologic conditions) or unable to perform baseline stress testing
* Scheduled for a coronary artery bypass graft (CABG) or a percutaneous transluminal coronary angioplasty (PTCA) procedure, or CABG procedure within 90 days or a PTCA procedure within 30 days of enrollment.
* Biventricular pacing system, or indication for Biventricular pacing system
* Myocardial infarction within 90 days of enrollment.
* Mechanical tricuspid or aortic valves.
* Ventricular assist device
* Prior heart transplant
* Pregnant or planning to become pregnant during the study
* Age below 18
* Subject participating in another study, unrelated to CCM, at the same time (or within 30 days prior to enrollment to this study)
* Subjects on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Comparison between the groups of the change in Peak VO2 from baseline to 24 weeks of follow-up. | from baseline to 24 weeks of follow-up

SECONDARY OUTCOMES:
Comparison of change in quality of life as measure (MLWHFQ), from baseline to 24 weeks of follow-up | from baseline to 24 weeks of follow-up
Comparison of change in NYHA class, from baseline to 24 weeks of follow-up | from baseline to 24 weeks of follow-up
Comparison of change in Peak VO2 from baseline to 24 weeks of follow-up for each of the following subgroups separately: Baseline EF <35% , baseline EF ≥35% | from baseline to 24 weeks of follow-up

OTHER OUTCOMES:
Comparison between the groups of the change in SHFM survival prediction model score from baseline to 24 weeks of follow-up | from baseline to 24 weeks of follow-up
Comparison between the groups of the change in MAGGIC survival prediction model score from baseline to 24 weeks of follow-up | from baseline to 24 weeks of follow-up
All-cause mortality | from baseline to 24 weeks of follow-up
Cardiovascular mortality | from baseline to 24 weeks of follow-up
Time to first event - cardiovascular related | from baseline to 24 weeks of follow-up
Time to first event - all causes | from baseline to 24 weeks of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, Prof., Principal Investigator — Herzzentrum Leipzig GmbH
Locations (8):
- Universitätsklinik Innere Medizin, Graz, Austria
- Germany (5):
  - Universtitätsklinikum; Medizinische Klinik I, Aachen
  - Universitätsklinikum; Kardiologie im Herzzentrum, Cologne
  - Helios Klinikum; 3. Medizinische Klinik, Erfurt
  - Albertinen Krankenhaus, Hamburg
  - Universität Leipzig; Abteilung für Kardiologie und Angiologie, Leipzig
- 4th Military Hospital, Wroclaw, Poland
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No